CLINICAL TRIAL: NCT03485677
Title: Open Label, Two Cohort (With and Without Imiglucerase), Multicenter Study to Evaluate Pharmacokinetics, Safety, and Efficacy of Eliglustat in Pediatric Patients With Gaucher Disease Type 1 and Type 3
Brief Title: Safety and Efficacy of Eliglustat With or Without Imiglucerase in Pediatric Patients With Gaucher Disease (GD) Type 1 and Type 3
Acronym: ELIKIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EFC13738; U1111-1172-2950 (Registry Identifier: ICTRP); 2024-510751-34 (Registry Identifier: CTIS); 2016-000301-37 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-04-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Gaucher's Disease Type I; Gaucher's Disease Type III
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat; imiglucerase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Eliglustat monotherapy (Experimental): Eliglustat for at least two years. Cohort 1 patients that experience significant clinical decline will receive rescue treatment.
  Rescue Treatment Step 1: Switch from eliglustat to imiglucerase monotherapy.
  Rescue Treatment Step 2: Patients who after 6 months of rescue therapy with imiglucerase monotherapy do not show improvement in the parameter(s) that led to the switch from eliglustat to imiglucerase, will then receive combination therapy with eliglustat + imiglucerase.
  Interventions: Drug: Eliglustat GZ385660
- Cohort 2: Eliglustat plus imiglucerase (Experimental): Eliglustat plus imiglucerase for three years, at the dose of enzyme replacement therapy received before enrollment. After Week 52, Cohort 2 patients will switch to eliglustat monotherapy for the remainder of the study if the desired clinical response has been achieved.
  Interventions: Drug: Eliglustat GZ385660; Drug: Imiglucerase GZ437843

INTERVENTIONS:
Drug: Eliglustat GZ385660 — Pharmaceutical form: Capsule, Liquid
  Route of administration: Oral
  Other Names: Cerdelga
Drug: Imiglucerase GZ437843 — Pharmaceutical form: Powder for solution for infusion
  Route of administration: Intravenous
  Other Names: Cerezyme
  Arms: Cohort 2: Eliglustat plus imiglucerase

SUMMARY:
Primary Objective:

Evaluate the safety and pharmacokinetics of eliglustat in pediatric patients (≥2 to <18 years old).

Secondary Objective:

Evaluate the efficacy of eliglustat and quality of life in pediatric patients (≥2 to <18 years old).

DETAILED DESCRIPTION:
The study will include a screening period of up to 60 days (Day -60 to -1), a primary analysis treatment period (Day 1 to Week 52), a long-term treatment period (Week 53 to Week 104), and an extension period continuing up to Week 364 (for patients who continue to demonstrate the clinical benefit from eliglustat monotherapy at Week 104). After study completion, patients will be encouraged to enroll in the International Collaborative Gaucher Group (ICGG) Gaucher Registry.

ELIGIBILITY:
Inclusion criteria :

* The patient is 2 to <18 years old at the time of informed consent.
* Male and female patients with a clinical diagnosis of Gaucher disease (GD) type 1 or type 3 with documented deficiency of acid beta-glucosidase activity by enzyme assay and glucocerebrosidase (GBA) genotype.
* Postmenarchal female patients must have a documented negative pregnancy test prior to enrollment and throughout the study. Patients must be willing to practice true abstinence in line with their preferred and usual lifestyle, or use a medically accepted form of contraception throughout the study.

Cohort 1 (Eliglustat monotherapy):

* Patients must have been receiving an enzyme replacement therapy (ERT) for a minimum of 24 months at a monthly dose equivalent to 30 U/kg to 130 U/kg of Cerezyme® (imiglucerase) with treatment ongoing at the time of enrollment. Patients must be at pre-specified treatment goals, as defined by:

  * Hemoglobin level for ages 2 to <12 years: ≥11.0 g/dL; for ages 12 to <18 years: ≥11.0 g/dL for females and ≥12.0 g/dL for males;
  * Platelet count ≥100,000/mm3;
  * Spleen volume <10.0 multiples of normal (MN);
  * Liver volume <1.5 MN;
  * Absence of GD related pulmonary disease, and severe bone disease, as defined below for Cohort 2.

Cohort 2 (Eliglustat plus imiglucerase):

* Patients must have been receiving an ERT for a minimum of 36 months at a dose equivalent to at least 60 U/kg of imiglucerase every 2 weeks, or at the maximum dose locally approved, at the time of enrollment with treatment ongoing at the time of enrollment and the dose stable for at least the 6 months preceding enrollment. Patients must have severe clinical manifestations of GD, as defined by the presence of at least one of the following:

  * GD related pulmonary disease such as interstitial lung disease (ILD). The diagnosis of ILD must be confirmed by the presence of reticulonodular densities on chest X-ray; AND/OR
  * Symptomatic bone disease characterized by pathological fracture, osteonecrosis, osteopenia/osteoporosis, or bone crisis occurring in the 12 months prior to enrollment; AND/OR
  * Persistent thrombocytopenia (<80,000/mm3) related to GD.

Exclusion criteria:

* Substrate reduction therapy for GD within 6 months prior to enrollment.
* Partial or total splenectomy if performed within 2 years prior to enrollment
* The patient is transfusion dependent, a history of esophageal varices or liver infarction, elevated liver enzymes, significant congenital cardiac defect, coronary artery disease or left sided heart failure; clinically significant arrhythmias or conduction defect such as Type 2 second degree or third degree atrioventricular (AV) block, complete bundle branch block, prolonged QTc interval, or sustained ventricular tachycardia (VT).
* The patient has any clinically significant disease other than GD.
* The patient has neurological symptoms other than oculomotor apraxia at study entry.
* The patient has received an investigational product within 30 days prior to enrollment.
* The patient is unable to receive treatment with imiglucerase due to a known hypersensitivity or is unwilling to receive imiglucerase treatment every 2 weeks.
* The patient has a known hereditary galactose intolerance, Lapp lactase deficiency or glucose galactose malabsorption, or is a CYP2D6 ultra-rapid metabolizer or indeterminate metabolizer.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetic (PK) parameter of eliglustat: Cmax | Weeks 2, 13, 26 and 52
  Maximum concentration (Cmax) of eliglustat in plasma
Assessment of PK parameter of eliglustat: AUC | Weeks 2 and 52
  Area under the plasma eliglustat concentration-time curve (AUC)
Adverse Events | Up to Week 364
  Number of adverse events in pediatric patients

SECONDARY OUTCOMES:
Change in hemoglobin level | Baseline and Week 52
  Absolute change from baseline for hemoglobin (g/dL) (Cohort 1 patients)
Change in platelet count | Baseline and Week 52
  Percent change from baseline for platelet count (Cohort 1 patients)
Change in liver volume | Baseline and Week 52
  Percent change from baseline for liver volume (Cohort 1 patients)
Change in spleen volume | Baseline and Week 52
  Percent change from baseline for spleen volume (Cohort 1 patients)
Pulmonary disease improvement | Baseline and Week 52
  Proportion of patients with improvement in pulmonary disease (Cohort 2 patients)
Bone disease improvement | Baseline and Week 52
  Proportion of patients with improvement in bone disease (Cohort 2 patients)
Thrombocytopenia | Baseline and Week 52
  Proportion of patients with improvement in thrombocytopenia (Cohort 2 patients)
Quality of Life | Baseline and Week 52
  Health-related quality of life will be measured by the Pediatric Quality of Life Inventory™ (PedsQL™) questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- Investigational Site Number : 0320001, Capital Federal, Buenos Aires, Argentina
- Canada (3):
  - Investigational Site Number : 1240002, Calgary, Alberta
  - Investigational Site Number : 1240003, Vancouver, British Columbia
  - Investigational Site Number : 1240001, Toronto, Ontario
- Investigational Site Number : 2500002, Bron, France
- Investigational Site Number : 3800002, Roma, Italy
- Japan (2):
  - Investigational Site Number : 3920002, Koshigaya-shi, Saitama
  - Investigational Site Number : 3920001, Minato-ku, Tokyo
- Russia (4):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430004, Moscow
  - Investigational Site Number : 6430005, Saint Petersburg
  - Investigational Site Number : 6430002, Tomsk
- Spain (3):
  - Investigational Site Number : 7240002, Barakaldo, Bizkaia
  - Investigational Site Number : 7240001, Esplugues de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240003, Zaragoza
- Sweden (2):
  - Investigational Site Number : 7520002, Gothenburg
  - Investigational Site Number : 7520001, Luleå
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920004, Adana
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920002, Izmir
- Investigational Site Number : 8260002, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC13738 Plain Language Results Summaries — https://www.trialsummaries.com/Study/StudyDetails?id=25745&tenant=MT_SNY_9011